CLINICAL TRIAL: NCT02106494
Title: A Phase 3 Clinical Study Protocol: A Prospective, Randomized, Placebo-Controlled, Double-Blind, Multicenter, Phase 3 Study of APF530 500 mg SC, Fosaprepitant 150 mg IV, and Dexamethasone vs. Ondansetron 0.15 mg/kg IV, Fosaprepitant 150 mg IV, and Dexamethasone for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Patients Receiving Highly Emetogenic Chemotherapy
Brief Title: A Prospective, Multicenter, Study of APF530 (Granisetron) SC for Prevention of CINV in Patients Receiving HEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2013-01
Record Dates: First submitted 2014-03-28; First posted 2014-04-08 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-10

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Highly emetogenic chemotherapy (HEC); Chemotherapy-Induced Nausea and Vomiting (CINV)
MeSH Terms: conditions — Vomiting | interventions — Granisetron; Ondansetron; fosaprepitant; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- APF530 500 mg SC (Experimental): APF530 500 mg (granisetron 10 mg) SC and ondansetron placebo IV (0.15 mg/kg) and fosaprepitant 150 mg IV and dexamethasone 12 mg IV on Day 1 of Cycle 1 in association with HEC
  Interventions: Drug: APF530; Drug: Ondansetron placebo; Drug: Fosaprepitant; Drug: Dexamethasone
- ondansetron 0.15 mg/kg IV (Active Comparator): Ondansetron 2 mg/mL solution to be administered at 0.15 mg/kg IV (up to a maximum of 16 mg) and APF530 placebo SC and fosaprepitant 150 mg IV and dexamethasone 12 mg IV on Day 1 of Cycle 1
  Interventions: Drug: Ondansetron; Drug: APF530 placebo; Drug: Fosaprepitant; Drug: Dexamethasone

INTERVENTIONS:
Drug: APF530
  Arms: APF530 500 mg SC
Drug: Ondansetron
  Arms: ondansetron 0.15 mg/kg IV
Drug: Ondansetron placebo
  Arms: APF530 500 mg SC
Drug: APF530 placebo
  Arms: ondansetron 0.15 mg/kg IV
Drug: Fosaprepitant
Drug: Dexamethasone

SUMMARY:
The primary study objective is to demonstrate the superiority of APF530 500 mg given subcutaneously (SC) compared with ondansetron 0.15 mg/kg given intravenously (IV) (up to a maximum of 16 mg) in the delayed-phase (> 24-120 hours) complete response (CR) rate (defined as no emesis and no use of rescue medications) in subjects receiving highly emetogenic chemotherapy (HEC) as defined by the 2011 ASCO CINV guidelines

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males or nonpregnant females who are 18-87 years of age at the time of enrollment.
* Subjects must have histologically or cytologically confirmed malignant disease.
* Subjects must be undergoing treatment with a HEC regimen according to the 2011 ASCO CINV guidelines for further details on the emetogenic classifications of chemotherapy agents for this study).
* A life expectancy > 6 months
* Subjects must be able to receive standardized doses of dexamethasone as required in the protocol for the prevention of emesis.
* Subjects must be characterized as having Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subjects must have adequate bone marrow, kidney, and liver function.
* Subjects must be able to swallow oral medications (pills) without difficulty.
* Subjects must be entering the first cycle of their current chemotherapy regimen.
* Subjects must be willing and able to comply with all testing and requirements defined in the protocol.
* Subjects must be able to provide voluntary, written, informed consent to participate in this study and must be able to fully understand the study requirements.
* Female subjects cannot be pregnant and must be adequately protected from conception for the duration of study, using at least one form of contraception. It is recommended that females and female partners of male subjects remain adequately protected from conception during the study and for up to 1 year following study participation.

Exclusion Criteria:

* Subject has a known hypersensitivity to granisetron or any 5-HT3 receptor antagonist.
* Subject has a history or presence of clinically significant abnormal 12-lead ECG or an ECG with QTc by Bazett's correction of > 450 msec in men and > 470 msec in women on the screening ECG.
* Subject has PR > 240 msec, QRS > 110 msec, or a history of prolongation of QT interval.
* Subject has a family history of long QT syndrome.
* Subject has a history of cardiac disease, including congenital long QT syndrome, angina, myocardial ischemia or infarction, congestive heart failure, myocarditis, or chest pain or dyspnea on exertion.
* Subject has an electrolyte disturbance, such as uncorrected hypokalemia/hyperkalemia, hypomagnesemia, or hypocalcemia.
* Subject has idiopathic cardiomyopathy, syncope, epilepsy, hypertrophic cardiomyopathy, or other clinically significant cardiac disease.
* Subject is pregnant or breast-feeding.
* Subject is planning to receive multiple-day chemotherapy.
* Subject has taken any of the following agents within 7 days prior to initiation of chemotherapy (the study): 5-HT3 receptor antagonists, phenothiazines, benzamides, domperidone, cannabinoids, or NK-1 receptor antagonist.
* Subject has taken any benzodiazepine within 1 day (24 hours) prior to initiation of chemotherapy (the study).
* Subject is scheduled to receive any other chemotherapeutic agent from Day 2 through Day 6.
* Subject is scheduled to receive any radiation therapy to the abdomen or pelvis from Day -5 through Day 6.
* Subject has received systemic corticosteroids or sedative antihistamines within 72 hours of Day 1 of the study, except as premedication for chemotherapy (e.g., taxanes, pemetrexed).
* Subject has symptomatic primary or metastatic central nervous system (CNS) disease.
* Subject has ongoing vomiting, retching, or nausea caused by any etiology, or has a history of anticipatory nausea and vomiting.
* Subject has vomited and/or has had dry heaves or retching within 24 hours prior to the start of HEC on Day 1.
* Subject is NOT able to swallow oral medications (pills) without difficulty.

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 942 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gelder, MD, Study Director — Heron Therapeutics
Locations (7):
- United States (7):
  - Arizona Oncology Associates, PC-HAL, Pheonix, Arizona
  - The Oncology Institute of Hope and Innovation, Downey, California
  - Compassionate Cancer Medical Center, Riverside, California
  - Northern Indiana Research, Mishawaka, Indiana
  - Northern Indiana Research, South Bend, Indiana
  - North Shore Oncology, East Setauket, New York
  - Gabrail Cancer Center Research, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schnadig ID, Agajanian R, Dakhil C, Gabrail NY, Smith RE Jr, Taylor C, Wilks ST, Schwartzberg LS, Cooper W, Mosier MC, Payne JY, Klepper MJ, Vacirca JL. APF530 (granisetron injection extended-release) in a three-drug regimen for delayed CINV in highly emetogenic chemotherapy. Future Oncol. 2016 Jun;12(12):1469-81. doi: 10.2217/fon-2016-0070. Epub 2016 Mar 21. PMID 26997579

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients receiving highly emetogenic chemotherapy were stratified by cisplatin and randomized 1:1 to one of two treatment arms
Groups:
- APF530 + Fosaprepitant + Dexamethasone: Day 1 - Single SC dose of APF530 500 mg (10 mg granisetron) + Placebo for Ondansetron IV+ Fosaprepitant 150 mg IV+ Dexamethasone 12 mg IV
  Day 2 - Dexamethasone 8 mg PO QD
  Days 3 and 4 - Dexamethasone 8 mg PO BID
- Ondansetron + Fosaprepitant + Dexamethasone: Day 1 - Single IV dose of Ondansetron 0.15 mg/kg (up to a maximum of 16 mg) + Placebo for APF530 SC+ Fosaprepitant 150 mg IV + Dexamethasone 12 mg IV
  Day 2 - Dexamethasone 8 mg PO QD
  Days 3 and 4 - Dexamethasone 8 mg PO BID
Period: Overall Study
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone
Started | 471 | 471
Safety Population | 456 | 459
Efficacy Population | 450 | 452
Completed | 445 | 446
Not Completed | 26 | 25

BASELINE CHARACTERISTICS:
Population: Patients with a histologically or cytologically confirmed cancer diagnosis were scheduled to receive first cycle single day highly emetogenic chemotherapy (HEC)
Groups:
- APF530 + Fosaprepitant + Dexamethasone: Day 1 - Single SC dose of APF530 500 mg (10 mg granisetron) + Placebo for ondansetron IV + Fosaprepitant 150 mg IV + Dexamethasone 12 mg IV
  Day 2 - Dexamethasone 8 mg PO QD
  Days 3 and 4 - Dexamethasone 8 mg PO BID
- Ondansetron + Fosaprepitant + Dexamethasone: Day 1 - Single IV dose of Ondansetron 0.15 mg/kg (up to a maximum of 16 mg) + Placebo for APF530 SC + Fosaprepitant 150 mg IV + Dexamethasone 12 mg IV
  Day 2 - Dexamethasone 8 mg PO QD
  Days 3 and 4 - Dexamethasone 8 mg PO BID
- Total: Total of all reporting groups
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone | Total
Number analyzed (Participants) | 450 | 452 | 902
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 333 | 334 | 667
  >=65 years | 117 | 118 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.74) | 55.6 (11.94) | 55.65 (11.84)
Gender [Count of Participants; unit: Participants]
  Female | 358 | 373 | 731
  Male | 92 | 79 | 171

OUTCOME MEASURES:

1. Primary Outcome: Delayed Phase Complete Response (CR) Rate
Description: Percentage of Participants with no emesis and no rescue medication in patients receiving HEC in the delayed phase (24 to 120 hours) of CINV.
Time Frame: 24 - 120 Hours
Population: Modified Intent to Treat (mITT) - all subjects in the randomized population who receive study drug and a HEC regimen and have post-baseline efficacy data.
Measure: Number; unit: percentage of participants
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone
Number analyzed (Participants) | 450 | 452
percentage of participants | 64.7 | 56.6

2. Secondary Outcome: Overall Complete Response Rate
Description: To determine the effect of APF530 on complete response rates in the overall phase (0 to 120 hours) of CINV.
Time Frame: 0 - 120 Hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone
Number analyzed (Participants) | 450 | 452
percentage of participants | 58.4 | 52.9

3. Secondary Outcome: Delayed Complete Control (CC) Rate
Description: To determine the effect of APF530 on complete control rates defined as no more than mild nausea, no emetic episodes [vomiting or retching], and no use of rescue medications in the delayed phase (24 to 120 hours) of CINV.
Time Frame: 24 - 120 Hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone
Number analyzed (Participants) | 450 | 452
percentage of participants | 60.7 | 53.1

4. Secondary Outcome: Overall Complete Control Rate
Description: To determine the effect of APF530 on complete control rates defined as no more than mild nausea, no emetic episodes [vomiting or retching], and no use of rescue medications in the overall phase (0 to 120 hours) of CINV.
Time Frame: 0 - 120 Hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone
Number analyzed (Participants) | 450 | 452
percentage of participants | 54.7 | 49.6

5. Secondary Outcome: Rate of No Emetic Episodes
Description: To determine the effect of APF530 on the rate of no emetic episodes (vomiting or retching) in the overall phase (0 to 120 hours) of CINV.
Time Frame: 0 - 120 Hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone
Number analyzed (Participants) | 450 | 452
percentage of participants | 82.2 | 79.2

ADVERSE EVENTS:
Time Frame: The reporting period for AEs was the period starting from the time of informed consent signature until 30±3 days after study drug administration (Day 1 of chemotherapy cycle). Treatment-emergent AEs were those that either began or increased in severity after administration of study drug and within 8 days of study drug administration.
Description: Events other than injection site reactions were collected by non-systematic assessment. Injection site reactions were also collected via patient diaries.
Arm/Group | APF530 + Fosaprepitant + Dexamethasone | Ondansetron + Fosaprepitant + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 42/456 | 28/459
Other Adverse Events (participants affected / at risk) | 411/456 | 407/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APF530 + Fosaprepitant + Dexamethasone (N=456) | Ondansetron + Fosaprepitant + Dexamethasone (N=459)
Febria Neutropenia (Blood and lymphatic system disorders) | 9 | 6
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Mouth Haemmorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Pyrexia (General disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Breast Abscess (Infections and infestations) | 0 | 1
Breast Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Injection Site Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Post procedural cellulitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1
Chemical Peritonitis (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Intracranial Hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Convulsion (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 2 | 3
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | APF530 + Fosaprepitant + Dexamethasone (N=456) | Ondansetron + Fosaprepitant + Dexamethasone (N=459)
Neutropenia (Blood and lymphatic system disorders) | 26 | 30
Constipation (Gastrointestinal disorders) | 99 | 70
Diarrhea (Gastrointestinal disorders) | 39 | 35
Dyspepsia (Gastrointestinal disorders) | 27 | 32
Nausea (Gastrointestinal disorders) | 75 | 71
Fatigue (General disorders) | 95 | 109
Injection site bruising (General disorders) | 191 | 154
Injection site erythema (General disorders) | 77 | 127
Injection site haemorrhage (General disorders) | 23 | 36
Injection site nodule (General disorders) | 82 | 45
Injection site pain (General disorders) | 141 | 163
Injection site swelling (General disorders) | 45 | 53
Decreased Appetite (Metabolism and nutrition disorders) | 24 | 23
Dizziness (Nervous system disorders) | 25 | 25
Headache (Nervous system disorders) | 56 | 82
Insomnia (Psychiatric disorders) | 21 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A period of 60 working days for presentational material and abstracts and 90 days for manuscripts is permitted for the sponsor's review. The sponsor can request modifications of any manuscript or other materials to be published or presented. The sponsor can also request additional time to obtain additional patent protection or take such other measures to establish and preserve its intellectual property and proprietary rights before publishing information from this trial.